CLINICAL TRIAL: NCT01524835
Title: Live Lung Donor Cross-sectional Cohort Study
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT RELIVE-05
Record Dates: First submitted 2012-01-31; First posted 2012-02-02 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Lung Transplantation
Keywords: Tissue Donors; Lung; Transplants; Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Live lung donors: Live lung donors who participated in donation from 1993 through 2006

SUMMARY:
This study will gather information on the long-term effects of donating a lung lobe on living donors.

DETAILED DESCRIPTION:
Over time, the number of patients on the lung transplant waiting list and the number of lung transplants performed have greatly increased. Unfortunately, the number of patients on the waiting list has outpaced the transplant rate, resulting in a significant number of deaths for patients on the waiting list.

Live lung donation has the potential to decrease wait time for lung transplants and the rate of death for those awaiting transplants. However, since live lung donation typically utilizes one lobe of lung from each of two donors, transplantation puts two donors at risk for adverse events. Although live lung donation began in the early 1990s, there is still a great lack of published and comprehensive, long-term studies, leaving the outcome of live lung donation unclear. This study will assess post-donation outcomes in live lung donors. Specifically, investigators will determine the effects of live lung donation on lung function, quality of life, morbidity, psychosocial status, satisfaction with live lung donation, and decision-making associated with live lung donation. Information obtained from this study will allow potential future live lung donors and the interested public to become better informed, and may also assist potential donors in their decision-making process regarding the procedure. Furthermore, positive study results could potentially reassure previous live organ donors about uncertainties concerning their future health.

There will be 369 participants recruited for this study based on live lung donations, which occurred from 1993 through 2006. Study coordinators will contact eligible participants inviting participants to the study and answering any questions. Participants will have the option to partially or completely refuse participation. Each consenting donor will complete a series of questionnaires via phone and mail. The questions address issues related to the donor's quality of life, morbidity, psychosocial status, satisfaction with live lung donation, and decision-making associated with live lung donation. The questionnaires will take about one hour to complete. The coordinator will offer assistance regarding questionnaire completion and return. At the end of the study, a final brief status update will be obtained via phone interview.

In addition to questionnaires, participants will also be asked to participate in spirometry testing. For consenting participants, spirometry testing will be scheduled at either the two study sites or an approved Pulmonary Function Laboratory. During the test, the participant will breathe in and out of a plastic tube while a machine measures the amount and flow of air the donor breathes in and out. If deemed appropriate, the participant will do this test again a few minutes after being given albuterol, a drug which aims to optimize lung function. Spirometry testing will last about an hour.

ELIGIBILITY:
Inclusion Criteria:

* Donated a lung at University of Southern California or Washington University between January 1, 1993 and December 31, 2006

Exclusion Criteria:

* For questionnaire testing: inability to comprehend and complete questionnaires (with assistance)
* For spirometry: self-reported pregnancy, inability to reproducibly perform, and contraindications
* For post-bronchodilator spirometry: allergy to albuterol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Live lung donors who participated in transplantation during 1993 through 2006
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2010-08; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Spirometric lung function | Measured at time of scheduled spirometry testing

SECONDARY OUTCOMES:
Quality of life | Throughout study
Morbidity | Throughout study
Psychosocial status, including anxiety and depression symptoms | Throughout study
Satisfaction with live lung donation | Throughout study
Decision-making associated with live lung donation | Throughout study
Representativeness of participating live lung donor study sample | Throughout study
Predictors of donor outcome and/or status | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Mark Barr, MD, Principal Investigator — University of Southern California; Roger Yusen, MD, MPH, Study Chair — Washington University School of Medicine
Locations (2):
- United States (2):
  - University of Southern California, Los Angeles, California
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- [Result] Yusen RD, Hong BA, Messersmith EE, Gillespie BW, Lopez BM, Brown KL, Odim J, Merion RM, Barr ML; RELIVE Study Group. Morbidity and mortality of live lung donation: results from the RELIVE study. Am J Transplant. 2014 Aug;14(8):1846-52. doi: 10.1111/ajt.12771. PMID 25039865
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait
- Available data/document: Individual Participant Data Set: SDY294 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY294 — ImmPort study identifier is SDY294
- Available data/document: Study Protocol: SDY294 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY294 — ImmPort study identifier is SDY294. The study protocol is available in the Design tab section.
- Available data/document: Study summary, -design, -demographics, -study files: SDY294 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY294 — ImmPort study identifier is SDY294